CLINICAL TRIAL: NCT00253253
Title: Long-Term Outcome in Congenital Undescended Testis After Surgical Treatment by Orchidopexy
Status: Completed | Type: Observational
Sponsor: Medical Center Alkmaar (Other)
Other Study IDs: P05.936L
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Undescended Testis
Keywords: orchidopexy, long-term outcome, congenital
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to determine the long-term outcome in congenital undescended testis after surgical treatment by orchidopexy and to what extent orchidopexy is the treatment for congenital undescended testis.

ELIGIBILITY:
Inclusion Criteria:

* The orchidopexy has taken place in the Medical Center Alkmaar between 1986-2004
* The indication concerned a congenital undescended testis
* It concerns a first orchidopexy to the concerning testis

Exclusion Criteria:

* Orchidopexy has taken place on an other reason than congenital undescended testis (for example: torsio testis)
* It concerns re-orchidopexy

Ages: 6 Months to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 181 (Actual)
Dates: Start 2006-08; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: W.W. M. Hack, MD, PhD, Study Director — Department of Pediatrics, Medical Centre Alkmar
Locations (1):
- Medical Center Alkmaar, Alkmaar, North Holland, Netherlands